CLINICAL TRIAL: NCT04559477
Title: Comparison of Static & Dynamic Back Extensor Endurance Exercises For Chronic Low Back Pain
Brief Title: Comparison of Static & Dynamic Back Extensor Endurance Exercises in LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00236 Ayesha Jamal
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Back Pain
Keywords: Low Back Pain; Endurance; Static; Dynamic; Exercises; Pain
MeSH Terms: conditions — Back Pain; Low Back Pain; Motor Activity; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static extension endurance exercise (Experimental): static back extension endurance exercise
  Interventions: Other: Static extension endurance exercise
- Dynamic extension endurance exercise (Active Comparator): dynamic back extension endurance exercise
  Interventions: Other: Dynamic extension endurance exercise

INTERVENTIONS:
Other: Static extension endurance exercise — Static extension endurance exercise were performed, 10 repetitions with 10 sec hold of each of exercises Heating pad:15 mins TENS: 15 mins
  35 min/session, 3 sessions/week for 6 weeks
  Arms: Static extension endurance exercise
Other: Dynamic extension endurance exercise — Dynamic extension endurance exercise with 10 repetitions of each of exercises which has been performed Heating pad:15 mins TENS: 15 mins
  35 min/session, 3 sessions/week for 6 weeks
  Arms: Dynamic extension endurance exercise

SUMMARY:
This study will help to find the effects of static and dynamic back extensors exercises for chronic low back pain.

DETAILED DESCRIPTION:
Low back pain (LBP) is a very common health problem worldwide and a major cause of disability which affecting performance at work and general well-being. Determine the effects of static and dynamic back extensors exercises for chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Females
* 25-55 years
* Low back pain > 3 month
* Postural dysfunction

Exclusion Criteria:

* Red flags indicative of serious spinal pathology with signs and symptoms of nerve root compromise (with at least two of dermatomal sensory loss, myotomal muscle weakness and reduced lower limb reflexes)
* Individuals with any obvious spinal deformity or neurological disease;
* Pregnancy
* Previous spinal surgery
* Previous experience of static and dynamic endurance exercise.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females are included in the study
Enrollment: 52 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Roland-Morris Disability Questionnaire | 6th week
  The Roland-Morris Questionnaire (RMQ) is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale.
  The RMQ is a 24-item patient-reported outcome measure that inquires about pain-related disability resulting from LBP. Items are scored 0 if left blank or 1 if endorsed, for a total RMQ score ranging from 0 to 24; higher scores represent higher levels of pain-related disability
Modified Biering-Sorensen test of Static Muscular Endurance (BSME) | 6th week
  The BSME is used to assess the static back endurance. During the test the participant lay down on the plinth in the prone position with the upper edge of the iliac crests aligned with the edge of the plinth with their hands held by their sides. The lower body is fixed to the plinth by two non elastic straps located around the pelvis and ankles. Horizontality in the test position is ensured by asking the participant to maintain contact between his/her back and a hanging weighted ball. Once a loss of contact for more than 10 seconds is noticed, the participant is encouraged once to immediately maintain contact again. Once the participant could not immediately correct or hold the position or claimed to be fatigued the test is terminated.
  This test is time based, as long as the patient hold the position
Repetitive Arch-Up Test (RAUT) | 6th week
  Repetitive Arch-Up Test (RAUT) is used to assess the static back endurance. During the test, the participant lay in a prone position on the plinth with the arms positioned along the sides. The iliac crest is positioned at the edge of the plinth. The lower body is fixed to the plinth by two nonelastic straps located around the pelvis and ankles. With the arms held along the sides touching the body, the subject was asked to flex the upper trunk downward to 45∘ as indicated by a board. The participant then raised the upper trunk upwards to the horizontal position followed by returning back downward to 45 degrees to complete a cycle. The repetition rate is one repetition per two to three seconds. Once the movement becomes jerky or nonsynchronous, or do not reach the horizontal level, the subject is encouraged once to immediately correct the motion again. The test is terminated once the participant could not go on with the tempo of the motion or reported fatigue or exhaustion.
Numeric Pain Rating Scale (NPRS) | 6th week
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of pain. '0' usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible
Oswestry Disability Index (ODI), | 6th week
  Oswestry Disability Index is used to assess pain-related disability in persons with low back pain (LBP). The (ODI) is calculated based on each score of the ODQ, which consists of ten items. Each of the ten items is scored from 0 to 5, and the total is added and multiplied by 2. Therefore, the ODI ranges from 0 to 100. A higher score on the ODI indicates a more severe disability caused by LBP

CONTACTS AND LOCATIONS:
Overall Officials: Nazish Rafique, MSPT, Principal Investigator — Riphah International University
Locations (1):
- District Headquater hospital, Mirpur Mathelo, Mirpur Azad Kashmir, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Allegri M, Montella S, Salici F, Valente A, Marchesini M, Compagnone C, Baciarello M, Manferdini ME, Fanelli G. Mechanisms of low back pain: a guide for diagnosis and therapy. F1000Res. 2016 Jun 28;5:F1000 Faculty Rev-1530. doi: 10.12688/f1000research.8105.2. eCollection 2016. PMID 27408698
- [Background] Mbada CE, Ayanniyi O, Ogunlade SO. Effect of static and dynamic back extensor muscles endurance exercise on pain intensity, activity limitation and participation restriction in patients with long-term mechanical low-back pain. Med Rehabil. 2011;15(3):11-20.
- [Background] Mbada CE, Ayanniyi O, Ogunlade SO, Orimolade EA, Oladiran AB, Ogundele AO. Influence of Mckenzie protocol and two modes of endurance exercises on health-related quality of life of patients with long-term mechanical low-back pain. Pan Afr Med J. 2014 Jan 18;17 Suppl 1(Suppl 1):5. doi: 10.11694/pamj.supp.2014.17.1.2950. eCollection 2014. PMID 24624241
- [Background] Tanvi A, Shalini G, Parul R, Gaurav S. Effect of proprioceptive neuromuscular facilitation program on muscle endurance, strength, pain, and functional performance in women with post-partum lumbo-pelvic pain. IOSR J Dent Med Sci. 2013;7:60-7.
- [Background] Doo YT, Eom WS. Effect of Short Term Static• Dynamic Lumbar Stability Exercise on the Trunk Muscles Strength and Endurance of Chronic Low Back Pain Female College Students in Their 20's. The Official Journal of the Korean Academy of Kinesiology. 2016 May 31;18(2):63-9.
- [Background] Mayer JM, Childs JD, Neilson BD, Chen H, Koppenhaver SL, Quillen WS. Effect of Lumbar Progressive Resistance Exercise on Lumbar Muscular Strength and Core Muscular Endurance in Soldiers. Mil Med. 2016 Nov;181(11):e1615-e1622. doi: 10.7205/MILMED-D-15-00543. PMID 27849497
- [Background] McCaffery M, Beebe A. The numeric pain rating scale instructions. InPain: Clinic Manual for Nursing Practice 1989. Mosby, St. Louis.
- [Background] Alcántara-Bumbiedro S, Flórez-García MT, Echávarri-Pérez C, García-Pérez F. Oswestry low back pain disability questionnaire. REHABILITACION-MADRID-. 2006;40(3):150.
- [Background] Grotle M, Brox JI, Vollestad NK. Cross-cultural adaptation of the Norwegian versions of the Roland-Morris Disability Questionnaire and the Oswestry Disability Index. J Rehabil Med. 2003 Sep;35(5):241-7. doi: 10.1080/16501970306094. PMID 14582557
- See also: BASIC EXERCISES FOR THE LOW BACK — http://uhs.berkeley.edu/sites/default/files/LowBackPain.pdf